CLINICAL TRIAL: NCT04007887
Title: Effect of an Adult Education Program on Cardiovascular Outcomes in Post-myocardial-infarction Patients
Acronym: EDUCATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Spyridon Deftereos, Associate Professor of Cardiology, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CARD EBD2369/12-05-2017
Record Dates: First submitted 2019-06-30; First posted 2019-07-05 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Post-MI patients attending an adult education program designed to inform and motivate them on how to best control cardiovascular risk factors as a means to offer optimized secondary prevention of cardiovascular events
  Interventions: Other: Adult education program
- Controls (No Intervention): Usual care for post-MI patients

INTERVENTIONS:
Other: Adult education program — A 10-hour program embodying major adult education principles, designed to achieve cognitive involvement of patients in their treatment
  Arms: Intervention

SUMMARY:
A non-MD-led adult education program consisting in 10 one-hour sessions designed to provide information and motivation will be offered to patients who have recently been hospitalized for acute myocardial infarction (STEMI and NSTEMI), regarding the management of their treatment and strategies to aggressively optimize control of cardiovascular risk factors..

The intervention arm will be compared to a control group of patients treated with usual care.

ELIGIBILITY:
Inclusion Criteria:

* History of acute ST-elevation myocardial infarction (STEMI) or non-ST-elevation myocardial infarction (NSTEMI), Type Ι, according to the 3rd Universal Definition of MI, within the preceding 6 weeks
* Absence of substantial cognitive dysfunction (Mini Mental State examination score ≥24)

Exclusion Criteria:

- Age >80 years or <18 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2017-10-15 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Time to death or myocardial infarction or cerebrovascular event or unplanned hospitalization for cardiovascular reasons | 24 months
  Time from randomization to the composite endpoint of death or myocardial infarction or cerebrovascular event or unplanned hospitalization for cardiovascular reasons

SECONDARY OUTCOMES:
MACCE | 24 months
  Major cardio-/cerebro-vascular events (cardiovascular death, myocardial infarction, cerebrovascular event)

OTHER OUTCOMES:
Change in LDL-chol | 12 months
  Change from baseline to 12 months in LDL-cholesterol concentration
Change in body-mass index | 12 months
  Change from baseline to 12 months in the body-mass index
Change in arterial pressure | 12 months
  Change from baseline to 12 months in systolic arterial pressure (the mean of 3 office measurements)

CONTACTS AND LOCATIONS:
Locations (1):
- Athens University Hospital Attikon, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Giannopoulos G, Karageorgiou S, Vrachatis D, Anagnostopoulos I, Kousta MS, Lakka E, Giotaki S, Raisakis K, Sianos G, Toutouzas K, Cleman M, Deftereos S. A stand-alone structured educational programme after myocardial infarction: a randomised study. Heart. 2021 Jun 11;107(13):1047-1053. doi: 10.1136/heartjnl-2020-318414. PMID 33483355